CLINICAL TRIAL: NCT00871520
Title: Prognosis in Palliative Therapy - a Prospective Study on Survival Prognostication in Advanced Stage Cancer Patients
Brief Title: Prognosis and Survival Estimates in Palliative Therapy
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: Pro-08
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Cancer
Keywords: Palliative Care; Predictive Value of Tests; Prospective Studies; Survival Analysis; Survival prediction
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Palliative Therapy: Patients referred to the oncology / radiation oncology departments for palliative therapy.
  Interventions: Other: no specific interventions

INTERVENTIONS:
Other: no specific interventions — There are no specific interventions in this observational study

SUMMARY:
The accuracy of clinical survival estimates is tested in comparison to objective prognostic scores.

DETAILED DESCRIPTION:
* At presentation a clinical survival estimate is obtained in each patient.
* Survival is also estimated using published prognostic scores in palliative care.
* Prognostic scores based on blood samples, general symptoms, complaints, and performance status are calculated and validated, respectively
* Each patient completes questionnaires on psychological distress
* Survival estimates are limited to 6 months.
* Each patient is followed for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* oncologic disease confirmed
* incurable locally advanced or metastatic disease
* palliative treatment intended
* age > 18
* able to understand the study protocol
* able to complete the forms with assistance if necessary

Exclusion Criteria:

* therapy with curative intent
* regular clinical follow-up visit without disease progression
* ongoing therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive unselected cancer patients referred for palliative treatment to one of the participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 612 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Gripp, Dr., Principal Investigator — Universtity Hospital Duesseldorf, Radiation Oncology Department
Locations (3):
- Germany (3):
  - University Hospital Duesseldorf, Radiation Oncology Dept., Düsseldorf, North Rhine-Westphalia
  - Sana Kliniken Duesseldorf Benrath, Düsseldorf, North Rhine-Westphalia
  - Sana Kliniken Duesseldorf Gerresheim, MVZ Onkologie, Düsseldorf, North Rhine-Westphalia

REFERENCES:
- [Background] Gripp S, Moeller S, Bolke E, Schmitt G, Matuschek C, Asgari S, Asgharzadeh F, Roth S, Budach W, Franz M, Willers R. Survival prediction in terminally ill cancer patients by clinical estimates, laboratory tests, and self-rated anxiety and depression. J Clin Oncol. 2007 Aug 1;25(22):3313-20. doi: 10.1200/JCO.2006.10.5411. PMID 17664480